CLINICAL TRIAL: NCT03210844
Title: The Clinical Outcomes After Mini-incision Direct Anterior Approach and Microposterior Approach for Total Hip Arthroplasty
Brief Title: The Clinical Outcomes After Direct Anterior Approach and Microposterior Approach for Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511088RINB
Record Dates: First submitted 2017-06-25; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Total Hip Arthroplasty
Keywords: total hip arthroplasty; direct anterior; posterior approach

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct anterior approach: For the DAA group, we used single-incision direct anterior approach with a standard operation table in J Arthroplasty. 2008 Oct;23(7 Suppl):64-8. Epub 2008/10/24. . The incision size was 6-10 cm depending on the body build of the patient. The acetabularreaming was performed with an offset hemispheric reamer and acetabular component was inserted underfluoroscopic guidance. Femoral broaching was performed using a double-offset broach handle.Fluoroscopy was used to check the positioning and filling of femoral stem, as well as leg lengths.
  Interventions: Procedure: Surgical approaches of total hip arthroplasty
- Microposterior approach: The incision size was 6 - 10 cm depending on the body build of the patient. The differences of our micro-PA from Dorr's techniques were: First, no excision of the anterosuperior capsule and medial inferior capsule because the senior author believe that preservation of these structures could help to maintain the postoperative stability of the THA. Second, after the gluteus minimus muscle was elevated from the superior capsule, a superior capsulomy starting from 12 o'clock direction of acetabulum in decubitus position was made. The hip capsule was then incised in 12-to- 6-o'clock downward direction and curved down around femoral neck under the other short external rotators. We preserved short external rotators except piriformis tendon. Third, the capsular incision was continued inferiorly following 12-to- 6-o'clock downward direction of acetabulum to the transverse acetabular ligament. The tube structure of original hip capsule was divided into anterior and posterior half leaflets.
  Interventions: Procedure: Surgical approaches of total hip arthroplasty

INTERVENTIONS:
Procedure: Surgical approaches of total hip arthroplasty — Surgical approaches of total hip arthroplasty

SUMMARY:
Background The direct anterior approach (DAA) and micro-posterior approach (micro-PA) for total hip arthroplasty (THA) become popular approaches due to their fast recovery and good clinical outcomes. However, little is known if DAA is superior to micro-PA in implant positioning and functional outcomes for THA patients.

Methods The investigators conducted a non-randomized comparative study to compare component positioning and clinical outcomes of the consecutive unilateral primary THA patients operated with DAA techniques and that of those operated with micro-PA techniques by a single surgeon. The investigators used DAA techniques with standard operation table and micro-PA techniques featuring indirect-contracture-releasing capsulotomy, preservation of short external rotators except piriformis and conjoint tendon, and tendon-to-bone capsulotendinous repair. The investigators used propensity-score matching analysis to compare the postoperative THA component positioning and clinical outcomes in DAA and micro-PA groups.

DETAILED DESCRIPTION:
The direct anterior approach (DAA) has become a popular approach for total hip arthroplasty (THA) recently because of its atraumatic intermuscular plane, less tissue damage, and faster recovery. Studies comparing DAA with standard lateral or posterior approach showed DAA THAs have better results. These better results of DAA included possible lower dislocation rate, less perioperative pain, shorter length of hospital stay, and better implant position. However, DAA is a technic-demanding approach which needs a longer learning curve, and may endanger lateral femoral cutaneous nerve. DAA may also incurs a higher complication rates in obese patients than other approaches. Similarly, the mini-incision posterior approach (mini-PA) has most of the above-mentioned advantages of DAA except atraumatic intermuscular plane. Comparing with standard posterior approach, the mini-PA resulted in better function scores, shorter length of hospital stay, reduced blood loss, comparable radiographic outcome and complication rates. More recently, the micro-posterior approach (micro-PA), which evolves from mini-PA but preserves short external rotators of the hip except for the piriformis or conjoined tendon and includes all advantages of mini-PA, has been introduced into clinical practice and gained excellent clinical results.

Both DAA and micro-PA have their own advantages and disadvantages. Because of the fast recovery, both DAA and mini-PA were successfully used in outpatient THA. Furthermore, supine positioning during DAA facilitates the use intraoperative fluoroscopy to improve component positioning, while mini-PA and micro-PA utilize lateral decubitus position and achieve the safe zone of Lewinnek in only 60% of cases for cup positioning. In the learning curve of DAA, despite of the muscle-sparing advantage, there may be high early revision rate of THA. Therefore, both DAA and micro-PA have their own enthusiasts. To our knowledge, there were no studies comparing the results of DAA THAs with micro-PA THAs. Thus The investigators conducted a single-surgeon propensity-score matching study to compare these two approaches. Our hypothesis is that DAA THAs may have better results than micro-PA THAs in component positions and other clinical outcomes. The purpose of this study were to compare (1) the radiographic component positions, (2) the clinical outcomes, such as length of hospital stay, operative time, blood loss, perioperative pain scale, dislocation rates, and functional scores between DAA and micro-PA for THA.

Methods The investigators conducted a non-randomized comparative study to compare component positioning and clinical outcomes of the unilateral primary THA patients with DAA techniques and those with micro-PA techniques. The investigators received approval from institutional review board in National Taiwan University Hospital. The investigators recruited consecutive patients receiving unilateral primary THAs performed by a single surgeon (the senior author) between October 2013 and September 2014. The eligibility criteria were patients with unilateral hip arthritis indicated for THA. The excluding criteria were patients with previous THAs or patients indicated for revision THAs. A total number of 141 patients were recruited. Twenty-six of the patients underwent THAs with DAA and 115 of the patients underwent THAs with micro-PA. The patient demographics was shown in table 1. All the patients were regularly follow-up at least 2 year in out-patient clinics. The investigators used Trilogy acetabular cup system and ML-taper femoral components (Zimmer Inc., Warsaw, IN, United States) in all patients.

Perioperative protocol and discharge criteria Pre-operative digital templating was performed by the senior with AGFA IMPAX Orthopaedic Tools (Agfa Healthcare, Mortsel, Belgium) for every patient. Multimodal analgesia protocol including preoperative, intraoperative and postoperative medications (pregabalin, tramadol, acetaminophen, and celecoxib) was used in every patient. Intra-operatively, the patients received local infiltration analgesia with periarticular injection of diluted ketorolac and levobupivacaine solution. Additional intramuscular morphine was given for pain relief. The discharge criteria included (1) ambulation for 30 meters with assistive devices, (2) the ability to go up and down stairs with assistive devices, and (3) no need for intravenous or intramuscular analgesics.

Clinical outcomes Estimated blood loss, operation time and length of hospital stay were obtained from the electronic medical records. The patients' hemoglobin level was checked routinely on the day before operation and on the first and second post-operative days. The investigators also calculated the decreased amount of hemoglobin level as a more objective parameter for blood loss. Visual analogue scale (VAS) was recorded 4 times a day by nurse practitioners during hospitalization. The mean VAS on the first, second and third post-operative days were used for analysis respectively. Besides, the morphine dosage during hospitalization also served as another parameter of pain intensity. In addition to chart review, Harris hip score, Oxford hip score (OHS), and EQ5d scores were obtained for outcome evaluation at 3 months, 6 months, and 2 years after operation.

Radiographic parameters The stem alignment, acetabular cup abduction, anteversion angles and leg-length discrepancy were measured on digital anteroposterior (AP) pelvic radiographs. The radiographs were all obtained using a standardized technique with supine position, leg internally rotated and x-ray beam centered on pubic symphysis. For stem alignment, the investigators obtained proximal femoral axis, which was the line connecting centers of femoral canal at the levels of stem tip and lesser trochanter, and the femoral stem axis, which was the line connecting centers of femoral stem at levels of 2 centimeters and 5 centimeters proximal to the stem tip. The angle between proximal femoral axis and femoral stem axis was measured and analyzed as the stem alignment. The cup anteversion angle and abduction angle were means measured using AGFA IMPAX Orthopaedic Tool (Agfa Healthcare, Mortsel, Belgium). The leg-length discrepancy was the distance between the two lines from each lesser trochanter parallel to the inter-teardrop line.

Statistical Analysis With presumed achieved proportion of safe zone of Lewinnek in DAA and mini-PA, a minimum of 21 patients in each group were required, with an assumed two-sided alpha level of 5% and a power of 80%. Using body mass index (BMI), age and gender as covariates, 1:1 (DAA : micro-PA) propensity score matching was done. All the following analysis were calculated before and after propensity-score matching. The investigators used Mann-Whitney U test for comparison of continuous data and Chi-square test for categorical data. P < 0.05 was considered statistically significant. The software for analysis was STATA (StataCorp LP, Texas, USA).

Source of Funding Funding source did not play any role in this investigation.

ELIGIBILITY:
patients with unilateral hip arthritis indicated for THA

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unilateral hip arthritis indicated for THA
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic component positions - femoral alignment | Postoperative 2 year
  femoral alignment - to measure the angle between the stem axis and proximal femur axis on X ray 3. Cup inclination angle
Radiographic component positions - Cup anteversion angle | Postoperative 2 year
  to measure the cup anteversio angle on the X ray
Radiographic component positions - Cup inclination angle | Postoperative 2 year
  to measure the cup inclination angle on the X ray

SECONDARY OUTCOMES:
Leg length control | Postoperative 2 year
  The difference of the distance of bilateral lesser trochanter to the inter-teardrop line
Perioperative pain intensity | postoperative 1st, 2nd and 3rd days
  The record of visual analog pain scale on postoperative 1st, 2nd and 3rd days
Morphine usage | postoperative 1st, 2nd and 3rd days
  The morphine dosage which was needed on postoperative 1st, 2nd and 3rd days
Functional outcomes - Oxford hip score | Postoperative 2 year
  The record of Oxford hip score
Functional outcomes - EQ5D score | Postoperative 2 year
  The record of EQ5D score
Functional outcomes - Harris hip score | Postoperative 2 year
  The record of Harris hip score
Length of hospital day | Postoperative 2 week
  The record of admission date and discharge date
Dislocation rate | Postoperative 2 year
  We reviewed the image and medical record and asked the patients for dislocation rate
Operative blood loss | 1 day (operation day)
  The record of operation note for blood loss
Perioperative blood loss | 3 day (from the day before operation to postoperative day 1)
  We reviewed the hemoglobin level one day before the operation day and on the postoperative day 1. The hemoglobin difference was the parameter for perioperative blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chen-Ti, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No